CLINICAL TRIAL: NCT05892614
Title: Randomized, Double-blind, Placebo-controlled Proof-of-Concept (PoC) Study to Evaluate the Efficacy, Safety, and Tolerability of Efzofitimod in Patients With Systemic Sclerosis (SSc)-Related Interstitial Lung Disease (ILD) (SSc-ILD)
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of Efzofitimod in Patients With Systemic Sclerosis (SSc)-Related Interstitial Lung Disease (ILD) (SSc-ILD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: aTyr Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATYR1923-C-005
Record Dates: First submitted 2023-05-12; First posted 2023-06-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Interstitial Lung Disease
Keywords: ILD; SSc-ILD; Interstitial Lung Disease; lung inflammation; fibrosis; pulmonary function; efzofitimod; systemic sclerosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Pneumonia; Fibrosis; Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- efzofitimod 450 mg (Experimental): Administered IV infusion
  Interventions: Drug: efzofitimod 450 mg
- efzofitimod 270 mg (Experimental): Administered IV infusion
  Interventions: Drug: efzofitimod 270 mg
- Placebo (Placebo Comparator): Administered IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: efzofitimod 450 mg — IV infusion over approximately 60 minutes every 4 weeks
  Arms: efzofitimod 450 mg
Drug: efzofitimod 270 mg — IV infusion over approximately 60 minutes every 4 weeks
  Arms: efzofitimod 270 mg
Drug: Placebo — IV infusion over approximately 60 minutes every 4 weeks
  Arms: Placebo

SUMMARY:
This is a 2-Part study with Part A, a double-blind, randomized, placebo-controlled, PoC study to evaluate the efficacy, safety, and tolerability of efzofitimod in patients with SSc-ILD. The primary objective of the study is to evaluate the PoC for efficacy in a population with SSc-ILD. While improvement of ILD is the outcome of interest, the study will also evaluate changes in the skin. After initial screening (up to 4 weeks), approximately 25 eligible participants will be randomized 2:2:1 to 1 of 2 active (experimental) dose arms or placebo, administered every 4 weeks up to and including Week 20. Part B is an optional open-label extension to Part A in which participants can receive 450 mg efzofitimod every 4 weeks for 6 doses.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SSc based on ACR/ EULAR criteria (2013)
2. Overall duration of SSc < 84 months from the first non-Raynaud symptom manifestation prior to Day 1
3. HRCT obtained at the Screening Visit or within the 3 months prior to Screening consistent with SSc-ILD (adjudicated by a central reader) AND with pulmonary involvement > 10%
4. Clinical presentation at Screening consistent with lcSSc (up to 40% of patients) or dcSSc
5. MMF of ≥ 2 gm/day (or equivalent doses of other mycophenolate based compounds) for 3 months prior to Day 1 OR When documented intolerance to mycophenolates (in discussion with the Medical Monitor): treatment with maximum tolerated dose of MMF is acceptable, if < 2 gm/day, provided the cumulative duration of dosing has exceeded 3 months, OR An adequate dose and duration of an alternate immunosuppressant with a stable dose for the 4 weeks prior to baseline is also allowed.

Exclusion Criteria:

1. Pulmonary disease with FVC %pred ≤ 45% OR DLco %pred ≤ 30%; FEV1/FVC ratio < 0.7
2. Participants with pulmonary artery hypertension on parenteral therapy or with clinical evidence of right heart failure
3. HRCT obtained in the 3 months prior to Screening consistent with other confounding pathology.
4. Treatment with corticosteroids (> 10 mg/day of prednisone or equivalent) within 2 weeks prior to Day 1
5. Treatment with more than 1 immunosuppressant (e.g., MMF, methotrexate [MTX], azathioprine [AZA], or leflunomide)
6. Any treatment in the 12 months prior to Day 1 with any of the following: rituximab, intravenous immune globulin (IVIG), tocilizumab, cyclophosphamide, pirfenidone, tyrosine-kinase inhibitors (e.g., imatinib, nilotinib, dasatinib)
7. Rheumatic autoimmune disease other than SSc, Is an active, heavy smoker of tobacco/nicotine-containing products
8. History of (anti-Jo-1) anti-synthetase syndrome or Jo-1 positive at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in forced vital capacity (FVC) in mL | 24 weeks
Annual rate of decline in FVC in mL | 24 weeks
Annual rate of decline in FVC in percent predicted | 24 weeks
Change in HRCT fibrosis score | Baseline to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carey, Study Director — aTyr Pharma, Inc.
Locations (13):
- United States (13):
  - aTyr Investigative Site, Los Angeles, California
  - aTyr Investigative Site, San Diego, California
  - aTyr Investigative Site, Miami, Florida
  - aTyr Investigative Site, Chicago, Illinois
  - aTyr Investigative Site, New Orleans, Louisiana
  - aTyr Investigative Site, New York, New York
  - aTyr Investigative Site, Cleveland, Ohio
  - aTyr Investigative Site, Oklahoma City, Oklahoma
  - aTyr Investigative Site, Charleston, South Carolina
  - aTyr Investigative Site, Dallas, Texas
  - aTyr Investigative Site, Houston, Texas
  - aTyr Investigative Site, Salt Lake City, Utah
  - aTyr Investigative Site, Richmond, Virginia